CLINICAL TRIAL: NCT05223361
Title: Cardiopulmonary Bypass Prime Solution in Patients Undergoing Heart Valve Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rajaie Cardiovascular Medical and Research Center (Other)
Collaborators: Heart Valve Disease Research Center (Unknown)
Responsible Party: Principal Investigator, Rajaie cardiovascular medical & research center, Rajaie Cardiovascular Medical and Research Center, Rajaie Cardiovascular Medical and Research Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: HVDRC-01
Record Dates: First submitted 2022-01-08; First posted 2022-02-03 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2022-01

CONDITIONS: Heart Valve Diseases
MeSH Terms: conditions — Heart Valve Diseases | interventions — Ringer's Lactate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hydroxy ethyl starch (HES) (Active Comparator): Six percent hydroxy ethyl starch 130/0.4 additive to ringer lactate as priming solution during CPB
  Interventions: Drug: Six percent hydroxy ethyl starch 130/0.4; Drug: Ringer lactate
- Ringer lactate (RL) (Active Comparator): Ringer lactate as priming solution during CPB
  Interventions: Drug: Ringer lactate

INTERVENTIONS:
Drug: Six percent hydroxy ethyl starch 130/0.4 — 6% HES 130/0.4 additive to ringer lactate as prime solution
  Arms: Hydroxy ethyl starch (HES)
Drug: Ringer lactate — Ringer lactate as prime solution

SUMMARY:
In this randomized clinical trial, patients with undergoing open heart valve surgery will be enrolled into the study. Participants will be divided into two groups based on the priming solution type. The first group will receive hydroxyethyl starch (HES) 130/0.4 additive to ringer lactate (RL) and the second group will be given only RL as priming solution. All patients will be observed closely during postoperative days. Through follow up, bleeding/coagulopathy, renal function, hepatic function, and cerebral oxygenation will be recorded in both groups.

DETAILED DESCRIPTION:
Cardiopulmonary bypass (CPB) pump is a device for circulating blood in the body while the heart is undergone surgery. For providing circulating volume in the body we need to add about 1.5 to 2 lit fluids as priming solution in the CPB pump. Some fluids mainly included crystalloids, colloids, starch, and gelatin in an only fluid or in a combined formula. During CPB time, the blood dilution is caused by adding prime solution into the circulating volume, and consequently it decreases blood viscosity. Moreover, in addition to a decrease in hematocrit level, coagulation factors and plasma proteins can dramatically decreased. These processes may lead to bleeding events and tissue hypoperfusion and organ damages. To decrease complications, some modalities such as adding colloids to crystalloids have been implemented. On the other hand, any regimen for priming solution has its shortcomings need to be considered based on patient condition and surgical issue.

In this double blinded randomized clinical trial study, we aimed to compare the the effects of six percent HES 130/0.4 and RL as priming solutions on coagulation factors, renal function, hepatic function, and cerebral oxygenation in patients undergoing open heart valve surgery.

ELIGIBILITY:
Inclusion Criteria:

patients who provided written informed consent and had no heart failure (LVEF >55%), no hepatic failure (defined as aspartate aminotransferase (AST) >40 mg/dL and/or alanine aminotransferase (ALT) >40 mg/dL), no prior history of cardiac surgery, serum creatinine <1.5 mg/dL, no episode of drug-induced acute kidney injury within preoperative 5 days, no severe carotid stenosis in both or one of them, no emergency valvular stenosis, no infective endocarditis, no severe right ventricular failure, no hemoglobin <10 mg/dL, no body mass index >40 kg/m2, no heparin-induced thrombocytopenia, no cancer, no severe pulmonary valve insufficiency, no pulmonary function test <65% before heart valve surgery

Exclusion Criteria:

included consent withdrawal by the patient or by his/her proxy, allergic reaction to the drugs, the aortic cross clamp time greater than 120 minutes, on-pump time greater than 150 minutes, the performance of the retrograde autologous priming.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Number of participants required blood transfusion | Up to discharge, an average of 8 days
  The volume of blood transfusion after heart valve surgery

SECONDARY OUTCOMES:
Number of participants died in hospital | Up to discharge, an average of 8 days
  Any cause of death after heart valve surgery
Duration of ventilation time | During ICU admission, an average of 2 days
  The duration ventilation time after heart valve surgery
ICU length of stay | During ICU admission, an average of 2 days
  The length of stay in intensive care unit
Hospital length of stay | During hospital admission, an average of 8 days
  The length of stay in hospital after heart valve surgery
Number of participants required chest tube drainage | During hospital admission, an average of 8 days
  The amount of drainage from chest tube after heart valve surgery
Number of participants required re-operation for bleeding | During hospital admission, an average of 8 days
  Re-operation due to excessive bleeding after heart valve surgery
Number of participants died in one month | One month after surgery
  Any cause of death within one month after heart valve surgery
Changes in hemoglobin concentration | Up to 48 hours after heart valve surgery
  Changes in hemoglobin after heart valve surgery
Changes in hematocrit concentration | Up to 48 hours after heart valve surgery
  Changes in hematocrit after heart valve surgery
Changes in serum lactate concentration | Up to 48 hours after heart valve surgery
  Changes in serum lactate after heart valve surgery
Changes in serum blood sugar concentration | Up to 48 hours after heart valve surgery
  Changes in serum blood sugar after heart valve surgery
Number of participants with acute kidney injury | Up to 48 hours after heart valve surgery
  The development of acute kidney injury after heart valve surgery
Changes in liver enzyme concentration | Up to 48 hours after heart valve surgery
  Changes in liver enzyme after heart valve surgery
Amount of cerebral hemispheres' oxygenation | During cardiopulmonary bypass time
  The amount of cerebral oxygenation measured by INVOS in both hemispheres
Changes in coagulation parameters | Up to 48 hours after heart valve surgery
  Changes in coagulation parameters after heart valve surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Rajaie CMRC, Tehran, Iran

IPD SHARING:
Plan to Share IPD: Undecided
We will decide per request.